CLINICAL TRIAL: NCT07385456
Title: Effects of FES Arm Cycling on Functional Ability and Strength in People With Spinal Cord Injury: A Feasibility Study
Brief Title: FES Arm Cycling on Functional Ability and Strength in People With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 347696
Record Dates: First submitted 2025-12-03; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI); Upper Limb Function
Keywords: Spinal cord injury (SCI); FES Arm cycling; Functional Electrical Stimulation (FES); Upper limb functional ability; Upper limb strength
MeSH Terms: conditions — Spinal Cord Injuries | interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Intervention Model Description: Cohort, Feasibility design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES Arm Cycling (Experimental): FES arm cycling applied for up to 30 minutes. The intervention will be conducted 3 times a week for 6 weeks.
  Interventions: Other: Functional electrical stimulation (FES) arm cycling

INTERVENTIONS:
Other: Functional electrical stimulation (FES) arm cycling — FES arm cycling 3 times a week for 6 weeks.

SUMMARY:
The goal of this feasibility study is to determine if Functional Electrical Stimulation (FES) arm cycling can be used to improve arm functional ability and arm strength in people with Spinal Cord Injury (SCI). The main questions it aims to answer are:

* What is the feasibility of FES UL cycling in people with acute tetraplegia?
* What are the potential effects of FES UL cycling on strength and functional ability in people with acute tetraplegia?

Participants will:

* Complete an FES arm cycling intervention 3 times a week for 6 weeks.
* Complete assessments for upper limb function and strength pre and post-intervention.
* Complete questionnaires about upper limb and overall function and quality of life, pre and post-intervention.

DETAILED DESCRIPTION:
All inpatients admitted to the Queen Elizabeth National Spinal Injuries Unit for initial inpatient rehabilitation following acute SCI who fulfil the inclusion criteria will be invited to take part in the current study. Throughout the intervention participants will receive usual care. Once informed consent is gained participant demographics will be recorded (sex, age, level of SCI and severity classified by the INSCSCI, mechanism of injury and time since injury). Following this baseline assessments of upper limb function, overall function and quality of life will be recorded using a series of assessments and questionnaires.

Once baseline assessments are completed setting up of the Functional Electrical Stimulation (FES) arm cycling will begin.

Each participant will be assigned an individual log-in and upper limb cycling program on the RT300 (Restorative Therapies) FES Stationary Cycling Bike based in the QENSIU. The first session will involve assessment of parameters for each muscle using the FES. Muscles that do not have antigravity function will be targeted for stimulation. Up to 12 upper limb muscles groups can be stimulated with the RT300 via electrodes on the skin in a coordinated cyclic motion. The skin will be checked to make sure there are no burns or wounds, then ensuring the skin is clear, the electrodes will be placed over the muscles. The muscles being stimulated will likely include anterior deltoid, posterior deltoid, biceps, triceps, wrist and finger extensors and / or wrist and finger flexors. Assessment of participant tolerance and appropriate parameters with the FES will involve 2 adhesive electrodes being placed on the skin over the target muscle and attached to the stimulator. The amplitude (intensity) of the stimulation will gradually be increased until a sufficient muscle contraction is observed, or the participant starts to experience discomfort, whichever comes first. Parameters will be manipulated to make the stimulation as comfortable as possible, but if a sufficient contraction can not be achieved within the patients comfort they will be withdrawn from the study. This will be repeated for each muscle on each arm, skin will be checked after each muscle. The maximum amplitude is 140mA. Pulse width will range from 150us to 450us depending on the muscle and frequency will be set at 40Hz. Once all muscle parameters have been identified, the participant will be set up on the arm ergometer with grip aids if required to maintain hand position on the handles while cycling. The speed of the ergometer will gradually be increased then the stimulation for all muscles will be gradually increased. The RT300 automatically stimulates the muscle at the point in the crank that the muscle would normally by active when cycling. A target of 2-3 minutes of arm cycling with stimulation will be set for the first session. The arm cycling measures are as follows: speed is measured in Revolutions per Minute (RPM) and will be set at 30 RPM for the first session. Resistance will initially be set at 0.5 Nm (Newton meters) but will be adjusted to help the participant to maintain the target cycling speed. The participant will be monitored for any adverse events throughout while FES arm cycling.

Following set up of the FES arm cycling, the intervention will begin consisting of 3 sessions a week for 6 weeks. An FES session will start with the electrode set up and amplitudes being set based on parameters determined during set up. There will be a 3-minute warm-up of arm cycling without FES. Stimulation will then be added for up to 30 minutes. The target speed will be set at 30 RPM and the participant will be encouraged to use their own efforts, assisted by the FES, to cycle at this speed. If the speed drops below 30 RPM, the resistance level will reduce and if required, a motor will activate to help maintain the target speed. A 2-minute cool down without the stimulation and resistance will finish the session. Rests can be taken as required during the cycling session but the session will be terminated if a participant needs to rests for any longer than 5 minutes, skin will also be checked every time the FES stimulation is stopped. Although a target of 30 minutes of FES application has been set, actual stimulation length for each session is tailored towards each participant and will be based on their tolerance to the FES which will be gradually built upon in the 6 weeks.

Once the 6 weeks are completed the same questionnaires and assessments will be completed with the addition of the participant's global impression of change questionnaire which will conclude the participants involvement in the intervention.

Feasibility will be measured throughout the intervention by recording recruitment rate and retention looking at the number of eligible participants and the number of participants recruited. The number of participants not enrolled and why, and the number of participants who drop-out and why.

Adherence will be recorded by the completion rates of the 6 week intervention (duration of the session and number of sessions and reasons for non-attendance at sessions).

Perceived burden/inconvenience/benefit will be reported by the participants using a questionnaire.

Safety of the intervention will be recorded if there are any adverse events or safety concerns. Any that occur due to the intervention will be determined by discussion between the research and clinical team.

Usual care will be reported by participants on a self recall of what they attended each week of physiotherapy and occupational therapy.

FES parameters will also be reported as to stimulation levels, power, revolutions per minute and distance cycled.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at QENSIU
* Cervical level SCI (C8 or above) both complete and incomplete of less than 1 year in duration
* Medically stable to engage in physical rehabilitation
* Able to maintain seated position in manual or electric wheelchair for 3-4 hours per day
* Upper Extremity Motor Score below 30/50 on the ISNCSCI

Exclusion Criteria:

* Under 18 years old
* Unable to understand English (written and spoken)
* Uncontrolled Autonomic Dysreflexia
* Uncontrolled epilepsy
* Pregnant
* Current cancer diagnosis
* Pacemaker in situ
* Any upper limb injuries that may prevent participation in upper limb cycling e.g. arm fracture or open wound
* Taking part in another rehabilitation SCI trial that involves training of the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | From enrollment to the end of the intervention at week 7
  Recruitment rate (%)

SECONDARY OUTCOMES:
Attrition | From enrolment to the end of treatment at 7 weeks
  Number of dropouts as a percentage of number of participants recruited
Adherence | From enrolment to the end of treatment at 7 weeks
  Adherence (%) to the number of intervention sessions
Adverse Events | From enrolment to the end of treatment at 7 weeks
  Safety of the intervention self report of any adverse events and serious adverse events.
Perceived burden | From enrolment to the end of treatment at 7 weeks
  Perceived burden/inconvenience/benefit 9 point likert scale higher score more burden.
Muscle Strength | From enrolment to the end of treatment at 7 weeks
  Handheld dynamometry (kg) of major muscle groups of the upper limb
Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) | From enrolment to the end of treatment at 7 weeks
  Hand Function, 0-188 higher score = more hand function.
Capabilities of Upper Extremity Questionnaire (CUE-Q) | Baseline (week 0) and after the intervention (week 7)
  Subjective capability with the upper limb and hand, 0-128 higher score = more hand function.
Spinal Cord Independence Measure III self report (SCIM III SR) | From enrolment to the end of treatment at 7 weeks
  Overall functional ability, 0 - 100 high score = greater perceived independence
Global impression of change | End of treatment at 7 weeks
  Completed by participant. 0-7 higher score = greater impression of change.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided